CLINICAL TRIAL: NCT04414111
Title: Highly Suppressive Treg as a Biomarker for Immunologically Relevant Delayed (DGF) and Slow (SGF) Graft Function After Kidney Transplantation
Brief Title: Highly Suppressive Treg in Delayed and Slow Graft Function After Kidney Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: Mid-America Transplant (Other)
Responsible Party: Principal Investigator, Henry B. Randall, MD, MBA, FACS, Professor of Surgery, St. Louis University
Other Study IDs: 30530
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: DGF; Kidney Transplant; Complications
Keywords: DGF; SGF; Acute rejection; Kidney transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipient: Kidney transplant recipient
  Interventions: Diagnostic Test: Highly suppressive Treg measurement

INTERVENTIONS:
Diagnostic Test: Highly suppressive Treg measurement — Circulating highly suppressive Treg measurement

SUMMARY:
Delayed/slow graft function is the most common complication after kidney transplantation with an incidence over 20% and is the result of ischemia-reperfusion injury. The increased use of marginal kidney grafts to palliate the organ shortage is leading to a continued rise in the incidence of delayed/slow graft function. Delayed/slow graft function, however, is associated with an increased risk of acute rejection and graft failure. There are currently no clinically accepted biomarkers and no specific treatments for delayed/slow graft function. Regulatory T cells are protective in ischemia-reperfusion injury and rejection by suppressing pathologic immune responses. We hypothesize that the pre-transplant measurement of highly suppressive regulatory T cell is an accurate biomarker for delayed/slow graft function and its immunologic consequences. Ultimately, marginal kidney graft allocation could be directed to regulatory T cell-robust recipients and regulatory T cell-directed therapies could decrease marginal kidney graft discards without increasing delayed/slow graft function or impacting outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Adult kidney transplant candidates immediately prior to their kidney transplant surgery

Exclusion Criteria:

* < 18 years old
* Active immunosuppressive drug use
* Hepatitis C
* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Delayed graft function | 1 week
  Delayed graft function defined as dialysis requirement within the first week after kidney transplant
Slow graft function | 24 hours
  Slow graft function defined as a serum creatinine drop of less than 20% in the first 24 hours after kidney transplant

SECONDARY OUTCOMES:
Acute rejection | 1 year
  Kidney allograft biopsy-proven acute rejection according to Banff criteria

CONTACTS AND LOCATIONS:
Overall Officials: Henry Randall, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Loma Linda University Health Transplantation Institute, San Bernardino, California
  - Saint Louis University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided